CLINICAL TRIAL: NCT05432622
Title: Treatment Patterns and Outcomes for Patients With Stage IIIA Melanoma Receiving Adjuvant Systemic Therapy in the US Community Oncology Setting
Brief Title: A Study of Treatment Patterns and Outcomes in Participants With Stage IIIA Melanoma Receiving Adjuvant Systemic Therapy
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA209-7PG
Record Dates: First submitted 2022-06-21; First posted 2022-06-27 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Melanoma
Keywords: Anti-programmed cell death protein 1 (PD-1); Watchful waiting
MeSH Terms: conditions — Melanoma; Parkinson Disease 4, Autosomal Dominant Lewy Body

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (4):
- Nivolumab Monotherapy: Participants who started adjuvant nivolumab
- Pembrolizumab Monotherapy: Participants who started adjuvant pembrolizumab
- Dabrafenib + Trametinib Combination Therapy: Participants who started adjuvant dabrafenib + trametinib combination therapy
- No Treatment of a Systemic Therapy: Participants with no systemic treatment during the study observation period until record of recurrence

SUMMARY:
The purpose of this study is to examine real-world data among participants with stage IIIa melanoma initiating nivolumab as adjuvant treatment in the community practice setting by utilizing patient data from the United States Oncology Network (USON) iKnowMed (iKM) electronic health records (EHR) database.

ELIGIBILITY:
Inclusion Criteria:

* Participants diagnosed with Stage IIIA melanoma during identification period
* Participants underwent sentinel lymph node biopsy (SLNB) (index-event) during identification period
* Participants with a complete surgical resection at or following SLNB during the identification period
* Participants received nivolumab, pembrolizumab or dabrafenib/trametinib as adjuvant therapy in USON post-index event during the identification period (i.e., within 12 weeks of SLNB/resection); or received no treatment during the index period
* Participants receiving care at a USON site utilizing the full EHR capacities of the iKM database at the time of treatment
* Participants with ≥2 visits within the USON during the observation period
* Participants ≥18 years of age at first clinical diagnosis of melanoma

Exclusion Criteria:

* Participants with a previous systemic therapy prior to index
* Participants with a diagnosis of ocular or uveal melanoma during the study period
* Participants with a previous nonmelanoma cancer without complete remission for more than 3 years prior to index
* Participants with mucosal or acral melanoma during the study period
* Participants with systemic use of glucocorticoids during at the initiation of adjuvant therapy
* Participants enrolled in a clinical trial at any time during the study period
* Participants with a diagnosis and receiving treatment for another malignancy during the study observation period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants diagnosed with stage IIIA melanoma receiving an adjuvant systemic treatment regimen in the USON iKM EHR database were identified.
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2019-12-19 (Actual); Primary Completion 2023-04-26 (Actual); Study Completion 2023-07-11 (Actual)

PRIMARY OUTCOMES:
Time to Treatment Discontinuation (TTD) | Up to 39 Months
Recurrence-free Survival (RFS) | Up to 39 Months

SECONDARY OUTCOMES:
Number of Participants with Treatment-related Adverse Events (AEs) | Up to 39 Months
Time to Next Treatment (TTNT) | Up to 39 Months
Number of Participants with Treatment-Related Hospitalizations | Up to 39 Months
Number of Participants with Emergency Department Visits | Up to 39 Months
Overall Survival (OS) | Up to 39 Months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, The Woodlands, Texas, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html